CLINICAL TRIAL: NCT03555669
Title: UNCPM 21609 Project SOAR Mental Health: Evaluation of the Impact of a Depression Treatment Program on Mental Health and HIV Care Outcomes in Malawi
Brief Title: Project SOAR-Mental Health Malawi: Depression and HIV Integration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-2834
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2019-06

CONDITIONS: Depression; HIV/AIDS
Keywords: Implementation Science; Malawi
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The investigators will employ a multiple baseline evaluation design in two clinics to evaluate the impact of depression treatment on HIV outcomes. Patients who screen positive for depression using PHQ-9 during the "pre" period will comprise the comparison group, while patients who screen positive during the "post" period will comprise the active group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening Phase (Pre) Group (No Intervention): Patients who screen positive on the PHQ-9 for depression during the "pre" period will comprise the comparison group. Participants will receive "standard of care" depression treatment at the providers discretion.
- Treatment Phase (Post) Group (Experimental): Patients who screen positive during on the PHQ-9 for depression during the "post" period will comprise the active group. Participants will receive the depression treatment intervention in the form of anti-depressants and/or problem solving therapy (PST) based on their PHQ-9 score.
  Interventions: Other: Depression Treatment

INTERVENTIONS:
Other: Depression Treatment — The depression treatment program combines measurement-based antidepressant treatment with PST with clinical response appropriate to the level of depressive severity. Patients scoring 0-4 on the PHQ-9, indicating no depression, receive no treatment. Patients scoring 5-9 on the PHQ-9, indicating mild depressive symptoms that likely are not a full major depressive episode, are offered PST. Patients scoring 10 or above on the PHQ-9, indicating moderate-to-severe depressive symptoms, are first offered anti-depressants. For this group, PST will be an alternative or augmentation option for those who do not tolerate or respond to antidepressant treatment. All patients' depressive severity is monitored with the option of modifying their treatment plan if their symptoms worsen or do not improve.
  Arms: Treatment Phase (Post) Group

SUMMARY:
Depression is highly prevalent among people living with HIV (PLHIV) in Malawi and elsewhere in sub-Saharan Africa (SSA). Besides its high prevalence, depression likely represents an important barrier to consistent HIV care engagement and long-term viral suppression. However, the potential for depression treatment to improve HIV care outcomes has received little attention in the region, in part because of limited mental health infrastructure. In this study, the investigators will evaluate the impact of a depression treatment program integrated within existing HIV clinics on depression response, retention in HIV care, and viral suppression. It is expected that this evaluation will yield important evidence on the impact of depression treatment integrated with HIV care for improving HIV care and mental health outcomes in Malawi.

DETAILED DESCRIPTION:
Study population:

The evaluation will abstract screening data for adult (≥18 years old) patients newly initiating antiretroviral therapy (ART) who are screened for depression at the two clinics before and after the integration of the depression treatment program, and additional treatment and outcome data for those patients who screen positive for depression.

Study Size:

Across the two clinics, the investigators expect to abstract depression screening data for approximately 2,300 patients. The investigators expect to abstract further treatment and outcome data for approximately 640 patients who screen positive for mild, moderate, or severe depression.

Study Duration:

Evaluation and dissemination activities will last two years.

Study Evaluation:

To evaluate the impact of the mental health treatment program on HIV care outcomes, the investigators will collect data on HIV appointment adherence and viral load at 6 months following ART initiation.

To evaluate the impact of the mental health treatment program on mental health outcomes the investigators will collect data on depression symptoms at baseline through 6 months following ART initiation.

Study Design Overview:

The study will employ a pre-post design in two HIV clinics in Lilongwe to evaluate the impact of integrating the depression treatment program within existing clinic operations on HIV and mental health outcomes. The investigators will use existing medical records and the depression patient registry maintained by the Ministry of Health-run clinics to abstract routinely collected clinical data. Using these data, the investigators will compare mental health and HIV outcomes before and after the integration of the depression treatment program. Depressive symptoms will be measured with the Patient Health Questionnaire 9 (PHQ-9). The PHQ-9 is a self-report questionnaire designed to assess depression through nine questions that come directly from the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) signs and symptoms of major depression. Additionally, the investigators will conduct short qualitative interviews with clinic and Ministry of Health staff about the integration of the depression screening and treatment program and with patients on their understanding of depression and satisfaction with depression screening and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* HIV-infected
* Newly initiating antiretroviral treatment at one of the program sites
* Screened for depression

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2082 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who are retained in care | 6 months after ART initiation
  Retention in care is defined as attending sufficient HIV appointments to maintain ART supply through the first 6 months on ART.
Proportion of participants who are virally suppressed | 6 months after ART initiation
  Viral suppression is defined as HIV RNA viral load of <1,000 copies/mL. Viral loads are measured approximately 6 months after ART initiation.

SECONDARY OUTCOMES:
Proportion of participants who achieve depression remission (PHQ-9 score less than 5) | 6 months after ART initiation
  Depression remission is defined as scoring less than 5 on the PHQ-9 approximately 6 months after ART initiation. The PHQ-9 is a self-report questionnaire designed to assess depression through nine questions that come directly from the DSM-IV signs and symptoms of major depression. The 9 items describe problems associated with depression, and participants must rate how often the patient has been bothered by the problems in the last 2 weeks on a 0-3 scale. The scores are summed for a total depression score, ranging from 0-27, with 0-4 being minimum and indicating no depressive symptoms, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression. Depressive symptoms will be measured with the PHQ-9 at baseline through approximately 6 months after ART initiation.
Proportion of scheduled ART visits attended | 6 months after ART initiation
  ART visit attendance is defined as attending scheduled ART appointments over the first 6 months on ART.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pence, PhD, MPH, Principal Investigator — UNC Gillings School of Global Public Health; Michael Udedi, MBA MPhil, Principal Investigator — Malawi Ministry of Health
Locations (2):
- Malawi (2):
  - Area 18 Clinic, Lilongwe
  - Area 25 Clinic, Lilongwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulisewa K, Minnick CE, Stockton MA, Gaynes BN, Hosseinipour MC, Mphonda S, Sansbury G, Udedi MM, Pence BW. The acceptability of antidepressant treatment in people living with HIV in Malawi: A patient perspective. Glob Public Health. 2023 Jan;18(1):2201327. doi: 10.1080/17441692.2023.2201327. PMID 37088107
- [Derived] Udedi M, Stockton MA, Kulisewa K, Hosseinipour MC, Gaynes BN, Mphonda SM, Pence BW. The effectiveness of depression management for improving HIV care outcomes in Malawi: protocol for a quasi-experimental study. BMC Public Health. 2019 Jun 26;19(1):827. doi: 10.1186/s12889-019-7132-3. PMID 31242877
- [Derived] Udedi M, Stockton MA, Kulisewa K, Hosseinipour MC, Gaynes BN, Mphonda SM, Mwagomba BM, Mazenga AC, Pence BW. Integrating depression management into HIV primary care in central Malawi: the implementation of a pilot capacity building program. BMC Health Serv Res. 2018 Jul 31;18(1):593. doi: 10.1186/s12913-018-3388-z. PMID 30064418